CLINICAL TRIAL: NCT05693389
Title: The Efficacy of Acceptance and Commitment Therapy on Impulsivity and Suicidality Among Clients With Bipolar Disorders: A Randomized Controlled Trial
Brief Title: Efficacy of Acceptance and Commitment Therapy on Impulsivity and Suicidality Among Clients With Bipolar Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, ayman el-ashry, lecturer at psychiatric nursing and mental health, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013620/64/9/2022
Record Dates: First submitted 2022-12-25; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Bipolar Disorder
Keywords: Acceptance and commitment therapy; Bipolar disorders; Impulsivity; Suicidality
MeSH Terms: conditions — Bipolar Disorder; Impulsive Behavior; Suicidal Ideation | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with bipolar disorder who will partaicpmg in acceptance and commitment therapy (Active Comparator): patients with bipolar disorder who will participate in acceptance and commitment therapy
  Interventions: Behavioral: acceptance and commitment therapy
- patients with bipolar disorder who will be under routine hospital care (Placebo Comparator): patients with bipolar disorder who will be under routine hospital care
  Interventions: Other: routine hospital care

INTERVENTIONS:
Behavioral: acceptance and commitment therapy — ACT attempts to encourage psychological flexibility, acceptance of one's own experiences, and dedication to behaviours that are consistent with one's own values. ACT therapies focus on six key processes to improve psychological flexibility: engagement with the present moment, acceptance, defusion, self as context, values clarification, and committed action.
  Arms: patients with bipolar disorder who will partaicpmg in acceptance and commitment therapy
Other: routine hospital care — the patients with bipolar disorders who receive routine pharmacological treatment
  Arms: patients with bipolar disorder who will be under routine hospital care

SUMMARY:
Psychiatric nurses face a huge challenge in predicting and preventing suicide behaviour in their patients with bipolar disorders, but it may also be one of the most accurate measures of how well their clinical care is working. In addition to, high impulsivity scores are associated with increased overall functional impairment, a higher number of episodes with early onset, and a higher number of past suicide attempts, as well as increased substance intake. Thus, this study aimed at evaluating the efficacy acceptance and commitment therapy on impulsivity and suicidality among bipolar clients.

research hypnosis

* Clients who engaged in acceptance and commitment therapy had less impulsivity than the control group.
* Clients who engaged in acceptance and commitment therapy had less suicidality than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Clients had to be at least 18 years old
* able to converse intelligibly and meaningfully
* read and write
* have an illness that hadn't lasted more than 10 years to assure the client's functionality
* ready to take part in the study.

Exclusion Criteria:

* Clients who demonstrated psychotic symptoms
* attended another group sessions
* were intoxicated or under the influence of alcohol
* had any comorbidity were excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Impulsivity | up to 16 weeks
  This questionnaire has 20 items that assess five aspects of impulsivity: positive eagerness, negative urgency, lack of perseverance, lack of premeditation, and sensation seeking. Each of the five aspects is evaluated using four items on a four-point Likert scales with anchors 1 (=Strongly agree) and 4 (=Strongly disagree). An elevated prevalence of impulsivity is reflected in higher scores.To create the Arabic S-UPPS-P, investigators had a professional translator translate the original S-UPPS-P's items from English into Arabic, and then back-translated into Arabic.
Suicide Ideation | up to 16 weeks
  BSSI is a 19-item scale that assesses the presence and intensity of suicidal thoughts in the week before examination. Each item is rated on an ordinal scale of 0 to 2, and the total score ranges from 0 to 38. Individuals respond to the first five things that are excerpted. If an individual replies positively to the fifth item (scores 1 and 2), he or she answers the remaining items; otherwise, the questionnaire is finished. There was no cut-off point utilised to classify the scores. As a result, for data analysis, investigators used overall scale scores.The more score increased, the more the client vulnerable to suicide.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strasser ES, Haffner P, Fiebig J, Quinlivan E, Adli M, Stamm TJ. Behavioral measures and self-report of impulsivity in bipolar disorder: no association between Stroop test and Barratt Impulsiveness Scale. Int J Bipolar Disord. 2016 Dec;4(1):16. doi: 10.1186/s40345-016-0057-1. Epub 2016 Aug 17. PMID 27530736
- [Background] Shahed, H., Ghadam, H., Taghva, A., Ebrahimi, M. R., Donyavi, V., & Ghasemzadeh, M. R. (2020). Effectiveness of Acceptance and Commitment Therapy in Reducing Symptoms of Anxiety , Depression , and Suicidal Ideation in Iranian Veterans Referred to a Military Psychiatric Hospital.
- [Background] Pankowski S, Adler M, Andersson G, Lindefors N, Svanborg C. Group acceptance and commitment therapy (ACT) for bipolar disorder and co-existing anxiety - an open pilot study. Cogn Behav Ther. 2017 Mar;46(2):114-128. doi: 10.1080/16506073.2016.1231218. Epub 2016 Sep 19. PMID 27647353
- [Background] Bteich G, Berbiche D, Khazaal Y. Validation of the short Arabic UPPS-P Impulsive Behavior Scale. BMC Psychiatry. 2017 Jul 6;17(1):244. doi: 10.1186/s12888-017-1407-y. PMID 28683772
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Derived] El-Sayed MM, Elhay ESA, Taha SM, Khedr MA, Mansour FSA, El-Ashry AM. Efficacy of acceptance and commitment therapy on impulsivity and suicidality among clients with bipolar disorders: a randomized control trial. BMC Nurs. 2023 Aug 17;22(1):271. doi: 10.1186/s12912-023-01443-1. PMID 37592290